CLINICAL TRIAL: NCT03304756
Title: Phase II Study of Neoadjuvant Treatment of Locally Advanced Breast Cancer Patients With the CAP Regimen
Brief Title: Study of Neoadjuvant Treatment of Locally Advanced Breast Cancer With CAP Regimen
Acronym: CAPneo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, José Bines, Oncologist, Instituto Nacional de Cancer, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prot 82-07
Record Dates: First submitted 2017-08-11; First posted 2017-10-09 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Triple Negative Breast Cancer Patients
Keywords: locally advanced breast cancer; triple negative; cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAP (Experimental): Cisplatin (50 mg/m2) in combination with doxorubicin (50 mg/m2) and cyclophosphamide (500 mg/m2) every 21 days and for a total of 6 cycles
  Interventions: Drug: CAP

INTERVENTIONS:
Drug: CAP — cisplatin (50 mg/m2) in combination with doxorubicin (50 mg/m2) and cyclophosphamide (500 mg/m2) every 21 days and for a total of 6 cycles

SUMMARY:
This is a single arm, single center, non-randomized, phase II trial of stage IIB/III TNBC. Patients received neoadjuvant chemotherapy with cisplatin (50 mg/m2) in combination with doxorubicin (50 mg/m2) and cyclophosphamide (500 mg/m2) every 21 days and for a total of 6 cycles. After surgery, adjuvant chemotherapy consisting of docetaxel (75 mg/m2) every 21 days was further provided for 4 cycles. Primary outcome was pathological complete response in the breast and axilla (pCR; ypT0ypN0). Secondary outcomes were safety, disease-free survival and overall survival.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single arm, single center, phase II clinical trial. Patients received neoadjuvant chemotherapy with cisplatin (50 mg/m2, intravenous [IV], day 1) in combination with doxorubicin (50 mg/m2, IV, day 1) and cyclophosphamide (500 mg/m2, IV, day 1) every 21 days and for a total of 6 cycles (CAP regimen). Subsequent mastectomy plus axillary lymph node dissection was performed. Pathological specimen was analyzed to assess tumor response in the breast and axilla. Adjuvant chemotherapy consisting of docetaxel (75 mg/m2, IV) every 21 days was further provided for 4 cycles. In case of tumor progression during neoadjuvant treatment, CAP was discontinued and additional local or systemic treatment was provided at the discretion of the investigator. The protocol was approved by the institutional review board of National Cancer Institute - Brazil. All patients provided written informed consent. The Brazilian Group of Breast Cancer Studies (GBECAM) and National Cancer Institute -Brazil were the academic sponsors and National Cancer Institute- Brazil was the funding source of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with locally advanced breast cancer (stages IIB, IIIA and IIIB), confirmed anatomopathologically, with hormonal receptors (Estrogen and / or progesterone) and ERBB2 negative to the immunohistochemical study pattern.
2. Presence of measurable disease according to RECIST criteria.
3. Staging with chest X-ray, abdominal ultrasound and bone scintigraphy Without evidence of metastatic disease. Capture in bone scintigraphy should be Evaluated by simple radiographs.
4. Performance Status (PS) of Eastern Cooperative Oncology Group (ECOG) ≤ 2.
5. Adequate haematological function, evidenced by higher hemoglobin level Than 9 g / dl, neutrophil count greater than 1,500 / mm 3 and platelet count greater than 100,000 / mm 3.
6. Adequate liver function, evidenced by bilirubin levels below 1.5 of normal values and liver enzyme levels less than 2.5 times normal.
7. Adequate renal function, evidenced by creatinine levels lower than 1.5 times normal value and / or estimated creatinine clearance (Cockroft) greater than 50 ml / min.
8. Preserved cardiac function assessed by Doppler echocardiography.
9. Socio-cultural ability to understand a clinical study and the need to Attend regularly for medical examinations and appointments.

Exclusion Criteria:

1. Patients with a history of previous neoplasia, except non melanoma skin cancer.
2. Previously treatment of breast cancer with surgery, chemotherapy or Hormone therapy.
3. Presence of metastatic disease
4. Concomitant malignant neoplasm (including contralateral breast).
5. Presence of uncontrolled heart, kidney or lung disease.
6. Presence of uncontrolled diabetes mellitus.
7. Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-12-15 (Actual); Primary Completion 2012-04-15 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 6 months
  Pathological complete response (pCR) assessed by the local pathology lab, and defined as the absence of tumor (invasive and/or in situ) both in the breast and axilla (ypT0 ypN0)

SECONDARY OUTCOMES:
Safety assessed according to NCI CTCAE | 5 years follow-up
  Safety was assessed according to NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 3.0.
Disease-free survival (DFS) | 5 years follow-up
  DFS was defined as time from surgery to disease recurrence or death from any cause
Overall survival (OS) | 5 years follow-up
  OS was defined as time from surgery to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: José Bines, Doctorate, Study Chair — Instituto Nacional de Cancer; Otto Metzger, Oncologist, Study Director — Medical oncologist in Boston, and affiliated with Dana-Farber Cancer Institute; José Bines, Doctorate, Principal Investigator — Instituto Nacional de Cancer

IPD SHARING:
Plan to Share IPD: Yes
All data from this study was monitored by the GBECAM (Brazilian Group of studies on breast cancer) and the protocol approved by the research ethics committee of the National Cancer Institute.
  The collected data are archived in the research center, available for consultation in individual clinical records by patients, in addition to the source documents and folders with all regulatory material of the study.
  We are in the process of finalizing a scientific paper, to be published in an international magazine, in order to disseminate the results of the study.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Ferreira AR, Metzger-Filho O, Sarmento RMB, Bines J. Neoadjuvant Treatment of Stage IIB/III Triple Negative Breast Cancer with Cyclophosphamide, Doxorubicin, and Cisplatin (CAP Regimen): A Single Arm, Single Center Phase II Study (GBECAM 2008/02). Front Oncol. 2018 Jan 24;7:329. doi: 10.3389/fonc.2017.00329. eCollection 2017. PMID 29416986